CLINICAL TRIAL: NCT02657408
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase I Trial in Healthy Male Current Smoker Subjects to Assess Pharmacodynamic Effects on Segmental Endotoxin Induced Inflammatory Response and Safety of 4 Weeks Oral Administration of BI 1026706
Brief Title: Clinical Trial to Assess Pharmacodynamic Effects on Segmental Endotoxin Induced Inflammatory Response of BI 1026706 Versus Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1320.17; 2015-001789-25 (EudraCT Number)
Record Dates: First submitted 2016-01-14; First posted 2016-01-15 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-04

CONDITIONS: Healthy

ARMS (2):
- BI 1026706 (Experimental)
  Interventions: Drug: BI 1026706
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1026706
  Arms: BI 1026706
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary and secondary objectives of the current study are the assessments of anti-inflammatory pharmacodynamic effects on segmental endotoxin induced inflammatory response after 4 weeks treatment with BI 1026706.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent consistent with ICH-Good Clinical Practice (GCP) guidelines and local legislation prior to participation in the trial.
* Healthy volunteers of both sex between 18 and 65 years (inclusive) of age, on the day of subject's signature of informed consent.
* Healthy subjects as assessed by the investigator, based on a screening examination including medical history, physical examination, vital signs (blood pressure, pulse rate, body temperature), 12-lead ECG, lung function and clinical laboratory results.
* Forced expiratory volume (FEV1) of >80% and FEV1/Forced vital capacity(fFVC) of >70% of the predicted normal value at screening
* Current smokers with a smoking history of at least 1 pack year and with at least 1 cigarette per day in the previous year
* BMI (Body mass index) range: >18.5 and < 29.9kg/m2.
* Negative urine drug screening.
* Negative breath alcohol test.
* Negative skin prick test (performed within the 12 months prior to study start or at study start)
* Females NOT of childbearing potential are defined as: Women who are postmenopausal (12 months with no menses without an alternative medical cause; in questionable cases a blood sample with simultaneous levels of FSH above 40 U/L and estradiol below 30 ng/L is confirmatory) or who are permanently sterilized (defined as hysterectomy, bilateral oophorectomy or bilateral salpingectomy).
* Further inclusion criteria apply

Exclusion criteria:

* History of any relevant lung disease (i.e. Chronic Obstructive Pulmonary Disease (COPD), asthma, chronic bronchitis, pulmonary fibrosis, pulmonary alveolar proteinosis (PAP), pneumocystis infection, active tuberculosis, silicosis or any other lung surfactant overproduction syndromes).
* Subjects with clinically relevant abnormal hematology, blood chemistry, or urinalysis at the screening visit
* Any finding of the medical examination (including blood pressure, pulse rate, body temperature and ECG) deviating from normal and of clinical relevance.
* Subjects with a history of any clinically significant cardiovascular, metabolic, renal (including renal stones), hepatic, gastrointestinal, hematological, dermatological, venereal, neurological, psychiatric or other major disorders.
* Subjects with a malignancy for which the subject has undergone resection, radiation therapy or chemotherapy within the last five years. Subjects with treated basal cell carcinoma or fully cured squamous cell carcinoma are allowed to participate.
* Subjects with previous surgery of the gastro-intestinal tract likely to affect drug absorption.
* History of relevant orthostatic hypotension, fainting spells or blackouts.
* Subjects with clinically relevant infection or known ongoing clinically relevant inflammatory process.
* History of relevant allergy/hypersensitivity including allergy to drug or its excipients or medications in line with bronchoscopy (bronchodilators, sedatives and local anesthetics).
* Subjects with a marked baseline prolongation of QT/QTcB interval (such as repeated demonstration of a QTcB interval >450 ms), or any other relevant ECG finding at screening visit (Visit 1) according to the investigator.
* Neutrophil blood count indicative of immunosuppression according to the investigator at screening visit (Visit 1).
* Subjects with previous surgeries that may have left ferromagnetic material in the body, ferromagnetic implants or pacemakers.
* Participation in another study with any investigational product within 2 months prior to screening or if screening occurs within 6 half-lives of intake of another investigational drug (whichever is greater).
* Male subjects who do not agree to minimize the risk of female partners becoming pregnant from the first dosing day until 3 months after the trial medication treatment has finished.
* Subjects who are committed to an institution by way of official or juridical order will not be enrolled in the trial.
* Receipt of live (attenuated) vaccine within the 4 weeks prior to screening or during the trial.
* Subject is assessed as unsuitable for inclusion by the investigator; for instance, because he is not considered able to understand and comply with study requirements or has a condition that would not allow safe participation in the study.
* For female subjects:

  * Positive pregnancy test at screening Visit 1, pregnancy or plans to become pregnant within 30 days after study completion
  * Lactation
* Further exclusion criteria apply

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Fraunhofer ITEM, Hanover, Germany

REFERENCES:
- [Derived] Gress C, Vogel-Claussen J, Badorrek P, Muller M, Hohl K, Konietzke M, Litzenburger T, Seibold W, Gupta A, Hohlfeld JM. The effect of bradykinin 1 receptor antagonist BI 1026706 on pulmonary inflammation after segmental lipopolysaccharide challenge in healthy smokers. Pulm Pharmacol Ther. 2023 Oct;82:102246. doi: 10.1016/j.pupt.2023.102246. Epub 2023 Aug 9. PMID 37562641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, placebo-controlled, double-blind, parallel-group study in a single trial center. In this study 57 healthy smoking subjects were entered and randomized. Subjects were allowed to rescreened twice based on investigator´s judgment with new informed consent & unique study subject number.
Pre-assignment Details: All subjects (Subjs) were screened for eligibility to participate in trial. Subjs attended specialist site to ensure that they (the Subjs) met all implemented inclusion/exclusion criteria. Subjs were not to be randomised to trial drug if any of specific entry criteria was violated.
Groups:
- Placebo: Subjects were orally treated with matching placebo as film-coated tablets twice daily in the morning and evening from beginning on Day 1 (Visit 2) until Day 28.
- BI 1026706: Subjects were orally treated with BI 1026706 as film-coated tablets 100 mg twice daily in the morning and evening from beginning on Day 1 (Visit 2) until Day 28.
Period: Overall Study
Arm/Group | Placebo | BI 1026706
Started | 28 | 29
Completed | 25 | 22
Not Completed | 3 | 7
Not completed — Adverse Event | 3 | 7

BASELINE CHARACTERISTICS:
Population: Treated set: The treated set included all subjects who were randomized and treated with at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 1026706 | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Treated Set
  Years | 32.4 (8.4) | 30.8 (5.4) | 31.6 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Treated set
  Participants
    Female | 0 | 0 | 0
    Male | 28 | 29 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Treated set
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 28 | 29 | 57
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — All subjects were white in this trial Population: Treated set
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 28 | 29 | 57
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Total neutrophil count [Mean (Standard Deviation); unit: cells*10^3/mL] — Total neutrophil count at baseline (Visit6) Population: Pharmacodynamic set (PDS): The pharmacodynamic set included all treated subjects who had evaluable cell counts for the primary or secondary endpoints 24 h after segmental LPS challenge.
  cells*10^3/mL
    number analyzed (Participants) | 24 | 22 | 46
    (all) | 2.79 (2.46) | 3.39 (4.13) | 3.07 (3.34)

OUTCOME MEASURES:

1. Primary Outcome: Total Cell Count of Neutrophils in Bronchoalveolar Lavage (BAL) Fluid After 24 Hours of the Segmental Lipopolysaccharide (LPS) Challenge
Description: Total cell count of neutrophils in Bronchoalveolar Lavage (BAL) fluid after 24 hours of the segmental Lipopolysaccharide (LPS) challenge.
  The adjusted geometric means (gMeans) are obtained by exponentiating the Least Square (LS) means obtained by fitting an Analysis of variance (ANOVA) model on the natural log transformed endpoint values, adjusted for treatment effect. Standard errors are derived using the delta method.
Time Frame: Day 29
Population: Pharmacodynamic set (PDS): The pharmacodynamic set included all treated subjects who had evaluable cell counts for the primary or secondary endpoints 24 h after segmental LPS challenge.
Measure: Geometric Mean (Standard Error); unit: cells*10^3/mililiter (mL)
Arm/Group | Placebo | BI 1026706
Number analyzed (Participants) | 24 | 22
cells*10^3/mililiter (mL) | 687.02 (109.315) | 872.61 (145.019)
Statistical Analysis 1: Comparison: Placebo vs BI 1026706; The statistical model used for the primary analysis of primary endpoints was an ANOVA model on the logarithmic scale. This model included the effect 'treatment'; Test type: Equivalence — confirmatory statistical hypothesis tested; p = 0.3043, ANOVA; Geometric mean ratio (%) = 1.27, 90% CI 2-sided [0.86 to 1.87]

2. Secondary Outcome: Differential Cell Count of Neutrophils in BAL Fluid 24 h After Segmental LPS Challenge.
Description: Differential cell count of neutrophils in BAL fluid 24 h after segmental LPS challenge.
  The adjusted geometric means (gMeans) are obtained by exponentiating the LS means obtained by fitting an ANOVA model on the natural log transformed endpoint values, adjusted for treatment effect. Standard errors are derived using the delta method.
Time Frame: Day 29
Population: PDS
Measure: Geometric Mean (Standard Error); unit: Percentage of neutrophils
Arm/Group | Placebo | BI 1026706
Number analyzed (Participants) | 24 | 22
Percentage of neutrophils | 54.83 (3.094) | 55.41 (3.266)
Statistical Analysis 1: Comparison: Placebo vs BI 1026706; The statistical model used for the analysis was an ANOVA model on the logarithmic scale. This model included the effect 'treatment'; Test type: Equivalence — No statistical hypothesis tested; Geometric mean ratio (%) = 1.01, 90% CI 2-sided [0.88 to 1.16]

3. Secondary Outcome: Total Cell Count of Eosinophil in BAL Fluid After 24 Hours of the Segmental LPS Challenge
Description: Total cell count of eosinophil in BAL fluid after 24 hours of the segmental LPS challenge.
  The adjusted geometric means (gMeans) are obtained by exponentiating the LS means obtained by fitting an ANOVA model on the natural log transformed endpoint values, adjusted for treatment effect. Standard errors are derived using the delta method.
Time Frame: Day 29
Population: PDS
Measure: Geometric Mean (Standard Error); unit: cells*10^3/mL
Arm/Group | Placebo | BI 1026706
Number analyzed (Participants) | 24 | 22
cells*10^3/mL | 6.95 (2.744) | 10.72 (4.420)
Statistical Analysis 1: Comparison: Placebo vs BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — No statistical hypothesis tested; Geometric mean ratio (%) = 1.54, 90% CI 2-sided [0.59 to 4.03]

4. Secondary Outcome: Differential Cell Count of Eosinophil in BAL Fluid 24 h After Segmental LPS Challenge.
Description: Differential cell count of eosinophil in BAL fluid 24 h after segmental LPS challenge.
  The adjusted geometric means (gMeans) are obtained by exponentiating the LS means obtained by fitting an ANOVA model on the natural log transformed endpoint values, adjusted for treatment effect. Standard errors are derived using the delta method.
Time Frame: Day 29
Population: PDS
Measure: Geometric Mean (Standard Error); unit: Percentage of eosinophil
Arm/Group | Placebo | BI 1026706
Number analyzed (Participants) | 24 | 22
Percentage of eosinophil | 0.55 (0.200) | 0.65 (0.246)
Statistical Analysis 1: Comparison: Placebo vs BI 1026706; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — No statistical hypothesis tested; Geometric mean ratio (%) = 1.17, 90% CI 2-sided [0.49 to 2.85]

5. Secondary Outcome: Total Cell Count of Monocyte in BAL Fluid After 24 Hours of the Segmental LPS Challenge
Description: Total cell count of monocyte in BAL fluid after 24 hours of the segmental LPS challenge.
  The adjusted geometric means (gMeans) are obtained by exponentiating the LS means obtained by fitting an ANOVA model on the natural log transformed endpoint values, adjusted for treatment effect. Standard errors are derived using the delta method. Monocyte cell count is the only cell count which was assessed by means of flow cytometry.
Time Frame: Day 29
Population: PDS
Measure: Geometric Mean (Standard Error); unit: cells*10^3/mL
Arm/Group | Placebo | BI 1026706
Number analyzed (Participants) | 24 | 22
cells*10^3/mL | 240.04 (34.306) | 310.79 (46.393)
Statistical Analysis 1: Comparison: Placebo vs BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — No statistical hypothesis tested; Geometric mean ratio (%) = 1.29, 90% CI 2-sided [0.91 to 1.83]

6. Secondary Outcome: Differential Cell Count of Monocyte in BAL Fluid 24 h After Segmental LPS Challenge.
Description: Differential cell count of monocyte (determined by flow cytometry) in BAL fluid 24 h after segmental LPS challenge.
  The adjusted geometric means (gMeans) are obtained by exponentiating the LS means obtained by fitting an ANOVA model on the natural log transformed endpoint values, adjusted for treatment effect. Standard errors are derived using the delta method.
  Monocyte cell count is the only cell count which was assessed by means of flow cytometry.
Time Frame: Day 29
Population: PDS
Measure: Geometric Mean (Standard Error); unit: Percentage of monocyte
Arm/Group | Placebo | BI 1026706
Number analyzed (Participants) | 24 | 22
Percentage of monocyte | 19.16 (1.058) | 19.73 (1.138)
Statistical Analysis 1: Comparison: Placebo vs BI 1026706; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — No statistical hypothesis tested; Geometric mean ratio (%) = 1.03, 90% CI 2-sided [0.90 to 1.18]

7. Secondary Outcome: Total Cell Count of Macrophage+Monocyte in BAL Fluid After 24 Hours of the Segmental LPS Challenge
Description: Total cell count of macrophage+monocyte BAL fluid after 24 hours of the segmental LPS challenge.
  The adjusted geometric means (gMeans) are obtained by exponentiating the LS means obtained by fitting an ANOVA model on the natural log transformed endpoint values, adjusted for treatment effect. Standard errors are derived using the delta method.
  Cytospin microscopy method cannot clearly differentiate between macrophages and monocytes, the total and differential cell count of macrophages and monocytes are presented together.
Time Frame: Day 29
Population: PDS
Measure: Geometric Mean (Standard Error); unit: cells*10^3/mL
Arm/Group | Placebo | BI 1026706
Number analyzed (Participants) | 24 | 22
cells*10^3/mL | 488.95 (52.417) | 575.43 (64.431)
Statistical Analysis 1: Comparison: Placebo vs BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — No statistical hypothesis tested; Geometric mean ratio (%) = 1.18, 90% CI 2-sided [0.91 to 1.53]

8. Secondary Outcome: Differential Cell Count of Macrophage+Monocyte in BAL Fluid 24 h After Segmental LPS Challenge.
Description: Differential cell count of macrophage+monocyte in BAL fluid 24 h after segmental LPS challenge.
  The adjusted geometric means (gMeans) are obtained by exponentiating the LS means obtained by fitting an ANOVA model on the natural log transformed endpoint values, adjusted for treatment effect. Standard errors are derived using the delta method.
  Cytospin microscopy method cannot clearly differentiate between macrophages and monocytes, the total and differential cell count of macrophages and monocytes are presented together.
Time Frame: Day 29
Population: PDS
Measure: Geometric Mean (Standard Error); unit: Percentage of macrophage+monocyte
Arm/Group | Placebo | BI 1026706
Number analyzed (Participants) | 24 | 22
Percentage of macrophage+monocyte | 39.03 (2.499) | 36.54 (2.444)
Statistical Analysis 1: Comparison: Placebo vs BI 1026706; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — No statistical hypothesis tested; Geometric mean ratio (%) = 0.94, 90% CI 2-sided [0.80 to 1.09]

9. Secondary Outcome: Total Cell Count of Lymphocyte in BAL After 24 Hours of the Segmental LPS Challenge
Description: Total cell count of lymphocyte after 24 hours of the segmental LPS challenge.
  The adjusted geometric means (gMeans) are obtained by exponentiating the LS means obtained by fitting an ANOVA model on the natural log transformed endpoint values, adjusted for treatment effect. Standard errors are derived using the delta method.
Time Frame: Day 29
Population: PDS
Measure: Geometric Mean (Standard Error); unit: cells*10^3/mL
Arm/Group | Placebo | BI 1026706
Number analyzed (Participants) | 24 | 22
cells*10^3/mL | 20.99 (3.976) | 16.91 (3.346)
Statistical Analysis 1: Comparison: Placebo vs BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — No statistical hypothesis tested; Geometric mean ratio (%) = 0.81, 90% CI 2-sided [0.51 to 1.28]

10. Secondary Outcome: Differential Cell Count of Lymphocyte in BAL Fluid 24 h After Segmental LPS Challenge.
Description: Differential cell count of lymphocyte in BAL fluid 24 h after segmental LPS challenge.
  The adjusted geometric means (gMeans) are obtained by exponentiating the LS means obtained by fitting an ANOVA model on the natural log transformed endpoint values, adjusted for treatment effect. Standard errors are derived using the delta method.
Time Frame: Day 29
Population: PDS
Measure: Geometric Mean (Standard Error); unit: Percentage of lymphocyte
Arm/Group | Placebo | BI 1026706
Number analyzed (Participants) | 24 | 22
Percentage of lymphocyte | 1.67 (0.283) | 1.07 (0.190)
Statistical Analysis 1: Comparison: Placebo vs BI 1026706; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — No statistical hypothesis tested; Geometric mean ratio (%) = 0.64, 90% CI 2-sided [0.43 to 0.97]

ADVERSE EVENTS:
Time Frame: From first dose administration of the study medication to 4 days after last drug administration; up to 35 days.
Arm/Group | Placebo | BI 1026706
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/28 | 1/29
Other Adverse Events (participants affected / at risk) | 21/28 | 18/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | BI 1026706 (N=29)
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | BI 1026706 (N=29)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 2
Pyrexia (General disorders) | 0 | 3
Lower respiratory tract infection (Infections and infestations) | 3 | 2
Respiratory tract infection (Infections and infestations) | 0 | 2
Rhinitis (Infections and infestations) | 0 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 5 | 6
Procedural complication (Injury, poisoning and procedural complications) | 3 | 3
Procedural headache (Injury, poisoning and procedural complications) | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Headache (Nervous system disorders) | 13 | 4
Agitation (Psychiatric disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT02657408/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT02657408/SAP_001.pdf